CLINICAL TRIAL: NCT04957069
Title: Comparison of Surgical Outcomes Between Avulsion Fracture of the Achilles Tendon and Conventional Achilles Tendon Rupture--a Retrospective Study
Brief Title: Comparison of Surgical Outcomes Between Avulsion Fracture of the AT and Conventional ATR--a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018040
Record Dates: First submitted 2021-06-25; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Avulsion Fracture of the Achilles Tendon; Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Avulsion fracture: avulsion fracture of the Achilles tendon
  Interventions: Procedure: fixation
- Rupture: Achilles tendon rupture
  Interventions: Procedure: primary repair

INTERVENTIONS:
Procedure: fixation — double row fixation with 3-4 wire anchors
  Groups: Avulsion fracture
Procedure: primary repair — end-to-end repair
  Groups: Rupture

SUMMARY:
To compare the surgical outcomes between avulsion fracture of the Achilles tendon and conventional Achilles tendon rupture, collected and analysed information of patients preoperatively and postoperatively.

DETAILED DESCRIPTION:
Include 30 patients with avulsion fracture of the Achilles tendon and 30 patients with Achilles tendon rupture underwent surgical treatment in our institute. Collect and evaluate MRI, VAS, AOFAS, and FFI score preoperatively and postoperatively. Finally explore the surgical outcomes between avulsion fracture of the AT and conventional ATR.

ELIGIBILITY:
Inclusion Criteria:

* patients with avulsion fracture of the Achilles tendon or Achilles tendon rupture

Exclusion Criteria:

* neuromuscular related diseases
* other injuries of ankle joint

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 2013 to 2017, patients with avulsion fracture of the Achilles tendon or Achilles tendon rupture that underwent surgical treatment in our institute.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
MOCART | one year after sugery
  MOCART is a scoring system to evaluate the repair effect of cartilage injury.The minimum and maximum values of MOCART are 100 and 0, respectively. And higher scores mean a better outcome.

SECONDARY OUTCOMES:
VAS | pre-surgery, one year after sugery
  The Visual Analogue Scale (VAS) is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced. This gives them the greatest freedom to choose their pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. The minimum and maximum values of VAS are 10 and 0, respectively. And higher scores mean a worse outcome.
AOFAS | pre-surgery, one year after sugery
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient (to assess sagittal motion, hindfoot motion, ankle-hindfoot stability and alignment of the ankle-hindfoot). The scale includes nine items that can be divided into three subscales (pain, function and alignment). The minimum and maximum values of AOFAS are 100 and 0, respectively. And higher scores mean a better outcome.
FFI | pre-surgery, one year after sugery
  A Foot Function Index (FFI) was developed to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales. Both total and sub-scale scores are produced. The FFI was examined for test-retest reliability, internal consistency, and construct and criterion validity. Each scale is from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it required help) .

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, MD, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Undecided